CLINICAL TRIAL: NCT02233764
Title: Effect of Iron- and Zinc-Biofortified Pearl Millet (ICTP8203-Fe) Consumption on Growth and Immunity in Children Aged 12-18 Months in India
Brief Title: Effect of Iron/Zinc-Biofortified Pearl Millet on Growth and Immunity in Children Aged 12-18 Months in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: SNDT Women's University (Other); St. John's Research Institute (Other); Center for the Study of Social Change (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB #: 1403004556
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Iron Deficiency; Zinc Deficiency
Keywords: iron; zinc; pearl millet; India; children; trial; randomized
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FeZnPM (Experimental): The FeZnPM arm will consume iron- and zinc-biofortified pearl millet (ICTP8203-Fe).
  Interventions: Other: FeZnPM
- CtrlPM (Active Comparator): The CtrlPM arm will consume conventional pearl millet three times per day, six days per week, for 9 months. Children are anticipated to consume 25-30 grams of the pearl millet at each feeding. The pearl millet will be prepared using a variety of recipes such as porridges, breads, and biscuits.
  Interventions: Other: CtrlPM

INTERVENTIONS:
Other: FeZnPM — Iron and zinc biofortified pearl millet will be consumed three times per day, six days per week, for 9 months. Children are anticipated to consume 25-30 grams of the pearl millet at each feeding. The pearl millet will be prepared using a variety of recipes such as porridges, breads, and biscuits.
  Other Names: biofortified pearl millet, bajra, ICTP8203-Fe
  Arms: FeZnPM
Other: CtrlPM — Conventional pearl millet will be consumed three times per day, six days per week, for 9 months. Children are anticipated to consume 25-30 grams of the pearl millet at each feeding. The pearl millet will be prepared using a variety of recipes such as porridges, breads, and biscuits.
  Other Names: bajra, pearl millet
  Arms: CtrlPM

SUMMARY:
In this study, iron- and zinc-biofortified pearl millet will be fed to young children in Mumbai, Maharashtra, India over a period of nine months to measure growth and immune function in comparison to children receiving non-biofortified pearl millet.

DETAILED DESCRIPTION:
Iron and zinc deficiency remain a major worldwide public health problem, especially in developing countries such as India. In this randomized study, 700 children aged 12-18 months from Mumbai, Maharashtra, India will be fed either iron and zinc biofortified pearl millet or control pearl millet three times per day, six days per week, for nine months. The goal of this study is to examine the effects of iron and zinc biofortified millet on immune function, growth, and cognitive function in this age group. The key outcome measures are biomarkers of iron and zinc status, growth, and immune function. Serum concentrations of hemoglobin, ferritin, serum transferrin receptor, and zinc will be assessed at enrollment (baseline), at an intermediate time point (midline; random serial sampling) and after 9 months of follow-up (endline). Additionally, we will measure concentrations of C-reactive protein (CRP) and alpha 1-acid glycoprotein (AGP), as iron and zinc biomarkers can be influenced by inflammation. To assess cognitive function in a subset, multiple specific aspects of memory, attention, and processing speed will be assessed. Higher-level, integrative cognitive abilities that require the coordination of multiple specific functions, such as problem-solving and exploratory behavior and global aspects of attention during free play with toys, will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months, 0 days to 18 months, 30 days (at time of screening/baseline visit)
* Hemoglobin ≥9 g/dL

Exclusion Criteria:

* Age less than 12 months, 0 days or older than 18 months, 30 days (at time of screening/baseline visit)
* Hemoglobin < 9 g/dL and/or hemoglobinopathy
* Presence of severe malnutrition according to Wellcome Classification (marasmus, marasmic kwashiorkor, kwashiorkor, weight-for-height z-score < -3)
* Prior diagnoses of HIV/AIDS or Tuberculosis, or Current diagnosis of HIV/AIDS, malaria, Dengue fever, Tuberculosis requiring >1 day hospitalization
* Children who do not have a caretaker to bring him/her to feeding center
* Possibility of migrating out of the slum dwelling for longer than 4 weeks
* Prior or current consumption of iron or zinc supplements in the past 1 year
* Any known dietary allergies

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Iron status | Midline serial assessment/sample between months 2-7
  Determined by serum ferritin, sTfR, and total body iron
Iron status | Endline (nine months)
  Determined by serum ferritin, sTfR, and total body iron
Physical growth | Midline serial assessment/sample between months 2-7
  As determined by length/height, weight, head circumference, and mid-upper arm circumference.
Physical growth | Endline (nine months)
  As determined by length/height, weight, head circumference, and mid-upper arm circumference.
Immune function | 1 Midline serial assessment/sample between months 2-7
  Measurement of T cell counts and vaccine response ELISA assays.
Immune function | Endline (nine months)
  Measurement of T cell counts and vaccine response ELISA assays.

OTHER OUTCOMES:
Cognitive function | Midline serial assessment/sample between months 2-7, in a subset
  Higher-level, integrative cognitive abilities that require the coordination of multiple specific functions, such as problem-solving and exploratory behavior and global aspects of attention during free play with toys, will be assessed.
Cognitive function | Endline (nine months) in a subset
  Higher-level, integrative cognitive abilities that require the coordination of multiple specific functions, such as problem-solving and exploratory behavior and global aspects of attention during free play with toys, will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Mehta, MBBS, ScD, Principal Investigator — Cornell University; Jere D. Haas, Ph.D., Principal Investigator — Cornell University; Julia L. Finkelstein, Sc.D., Principal Investigator — Cornell University; Richard L. Canfield, Ph.D., Principal Investigator — Cornell University; Shobha Udipi, Ph.D., Principal Investigator — SNDT Women's University; Padmini Ghugre, Principal Investigator — SNDT Women's University; R. Potdar, Principal Investigator — Centre for the Study of Social Change-Mumbai; Anura Kurpad, Principal Investigator — St. John's Research Institute
Locations (3):
- India (3):
  - Centre for the Study of Social Change-Mumbai, Mumbai, Maharashtra
  - St. John's Research Institute, Karnataka
  - S.N.D.T. Women's University, Mumbai

REFERENCES:
- [Derived] Mehta S, Huey SL, Ghugre PS, Potdar RD, Venkatramanan S, Krisher JT, Ruth CJ, Chopra HV, Thorat A, Thakker V, Johnson L, Powis L, Raveendran Y, Haas JD, Finkelstein JL, Udipi SA; Project Sabal. A randomized trial of iron- and zinc-biofortified pearl millet-based complementary feeding in children aged 12 to 18 months living in urban slums. Clin Nutr. 2022 Apr;41(4):937-947. doi: 10.1016/j.clnu.2022.02.014. Epub 2022 Feb 24. PMID 35299084
- [Derived] Huey SL, Finkelstein JL, Venkatramanan S, Udipi SA, Ghugre P, Thakker V, Thorat A, Potdar RD, Chopra HV, Kurpad AV, Haas JD, Mehta S. Prevalence and Correlates of Undernutrition in Young Children Living in Urban Slums of Mumbai, India: A Cross Sectional Study. Front Public Health. 2019 Jul 12;7:191. doi: 10.3389/fpubh.2019.00191. eCollection 2019. PMID 31355176
- [Derived] Mehta S, Finkelstein JL, Venkatramanan S, Huey SL, Udipi SA, Ghugre P, Ruth C, Canfield RL, Kurpad AV, Potdar RD, Haas JD. Effect of iron and zinc-biofortified pearl millet consumption on growth and immune competence in children aged 12-18 months in India: study protocol for a randomised controlled trial. BMJ Open. 2017 Nov 14;7(11):e017631. doi: 10.1136/bmjopen-2017-017631. PMID 29138201
- [Derived] Huey SL, Venkatramanan S, Udipi SA, Finkelstein JL, Ghugre P, Haas JD, Thakker V, Thorat A, Salvi A, Kurpad AV, Mehta S. Acceptability of Iron- and Zinc-Biofortified Pearl Millet (Dhanashakti)-Based [corrected] Complementary Foods among Children in an Urban Slum of Mumbai, India. Front Nutr. 2017 Aug 25;4:39. doi: 10.3389/fnut.2017.00039. eCollection 2017. PMID 28971097